CLINICAL TRIAL: NCT03906565
Title: Open, Multicenter, Monotherapy, Phase II Clinical Study of Utidelone Injection in Patients With Advanced or Metastatic Colorectal Cancer After Failure or Intolerability to Second-line Standard Treatment
Brief Title: Clinical Study of Utidelone Injection in Patients With Advanced or Metastatic Colorectal Cancer
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The efficacy evaluation (based on current data) deviated too much from results of previous clinical trials. It's assumed that high dropout rate of subjects, mainly due to covid-19 epidemic in China in the past 3 years, is the main reason.
Sponsor: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Chengdu Biostar Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BG01-1811
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Advanced or Metastatic CRC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- utidelone (Experimental): Utidelone Injection: 40 mg/m2/day, IV transfusing over 90 min. on day 1-day 5 of each 21 day cycle, administered to enrolled patients with advanced or metastatic CRC
  Interventions: Drug: utidelone injection

INTERVENTIONS:
Drug: utidelone injection — utidelone monotherapy in patients with advanced or metastatic CRC by iv transfusing utidelone injection
  Other Names: UTD1 injection

SUMMARY:
To assess the effectiveness and safety of utidelone injection in patients with advanced or metastatic colorectal cancer (CRC) as a phase II trial

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form; good compliance during the whole study;
2. Histologically or cytologically confirmed diagnosis of unresectable advanced or metastatic CRC, not including appendix and anal canal cancer;
3. patients failed or intolerable to previous standard second-line treatment for locally advanced or metastatic CRC;
4. Patients who have not received previous bevacizumab therapy can be treated in combination with bevacizumab;
5. Patients who did not receive chemotherapy, radiotherapy, surgical therapy, molecularly targeted drug therapy 4 weeks prior to enrollment, with no plan for concurrent other chemotherapy and surgery;
6. Age 18 -70 years old, ECOG performance status of 0-2; Life expectancy≥ 3 months;
7. Patients must have at least one measurable target lesion with long axis ≥10 mm on CT or MRI, with short axis ≥15mm for lymph node based on RECIST 1.1, within 4 weeks before enrolment;
8. Seven days prior to treatment, haematology test should meet the following requirements (no treatment with G-CSF or TPO 14 days before test): HGB ≥90 g/L, ANC ≥1.5×109/L, PLT ≥100×109/L, WBC ≥3.0×109/L bilirubin ≤1.5×ULN, aspartate transaminase (AST)/ alanine transaminase (ALT) ≤2.5 ×ULN (patients with liver metastasis ≤5xULN), and creatinine clearance ≥50 mL/min;
9. Peripheral neuropathy (PN) ≤grade 1 on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 within 4 weeks before enrolment; patients with any grade of alopecia are eligible for enrolment;
10. Patients with no major organ dysfunctions and heart disease;
11. Women and men of childbearing potential must agree to take effective contraceptive measures during the study and within six months after the last treatment. Female patients must have negative urinary pregnancy test within 7 days before the first treatmment (postmenopausal women must have no menstruation for at least 12 months before they are considered unable to conceive);
12. Patients must agree to provide blood samples for specific biomarkers study;
13. No other concurrent investigational agents during the study.

Exclusion Criteria:

1. Patients having history of other malignancies except CRC within the last five years, but patients with fully recovered in situ cervix carcinoma or non-melanoma skin cancer are eligible;
2. No other anticancer therapies, such as chemotherapy, hormonal therapy, immunotherapy, antibody therapy and radiotherapy, or concurrent other chemotherapy during treatment;
3. Patients with uncontrollable brain metastasis, uncontrollable bone metastasis or recent risk of fracture;
4. Arterial or venous thrombosis or embolic events such as cerebrovascular accident (including TIA), deep venous thrombosis or pulmonary embolism occurred within one year;
5. history of symptomatic heart disease (including unstable angina, myocardial infarction and heart failure);
6. history of interstitial lung disease (ILD), such as interstitial pneumonia, pulmonary fibrosis, or evidence of ILD on baseline chest CT or MRI;
7. Patients with gastrointestinal bleeding, active gastrointestinal ulcer or gastrointestinal obstruction (including paralytic intestinal obstruction). Patients with gastrointestinal perforation or gastrointestinal fistula and abdominal abscess within 6 month;
8. Previous partial or total gastrectomy, or major operations (such as laparotomy, thoracotomy and intestinal resection) within 4 weeks；
9. Patients with AEs caused by any previous treatment (including systemic and local treatment) that have not yet restored to GRADE 1 (excluding hair loss);
10. Patients who are pregnanct (positive pregnancy test), breastfeeding or unwilling to take contraceptive measures during the trial;
11. active or uncontrollable infections requiring systemic treatment (except simple urinary or upper respiratory infections) within 2 weeks;
12. Severely allergic to Cremophor or having severe adverse events associated with paclitaxel in the past;
13. Patients with active pulmonary tuberculosis.Patients having obvious cough blood or hemoptysis of half a teaspoon (2.5 ml) or more during the last one month;
14. Existence of uncontrolled diabetes, hypertension, active or uncontrollable infections;
15. Patients with serous effusion (such as pleural effusion, pericardial effusion and ascites) with clinical symptoms requiring intervention or stabilization for less than 4 weeks;
16. Patients with radiology findings that tumors have invaded important perivascular areas or tumors that are highly likely to invade important blood vessels during treatments which may lead to fatal massive hemorrhage determined by investigators;
17. Patients with abnormal coagulation function and tendency to bleed;
18. Patients with known HIV infection or untreated active hepatitis B or C;
19. Patients with alcohol or drug addiction, or a history of uncontrollable mental illness, lack of or limited legal capacity;
20. Patients with other conditions determined by investigators that may affect compliance with study protocol and study evaluation and are not suitable for participating in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response to utidelone treatment | 6 months from first study treatment
  Reflected by percentage of tumor size reduction or regression, assessed by imaging techniques and expressed as Objective Response Rate (ORR）ORR is defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) according to RECIST. 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 1 year from first study treatment
  PFS is defined as the duration of time from first study treatment to disease progression or death from any cause as documented by the investigator
Overall survival (OS) | 2 year from first study treatment
  OS is defined as the duration of time from first study treatment until death from any cause.
Safety profile associated with utidelone injection | 1 year from first study treatment
  Observe and record adverse effects and severe adverse effects associated with utidelone injection

CONTACTS AND LOCATIONS:
Overall Officials: RUIHUA XU, MD, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Tianjin People's Hospital, Tianjin